CLINICAL TRIAL: NCT01607086
Title: A Randomised, Double-blind Study in Healthy Volunteers to Compare the Properties and Characteristics of an Investigational Formulation of Lamotrigine With Placebo
Brief Title: Compare the Properties and Characteristics of an Investigational Formulation of Lamotrigine With Placebo
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 111649
Record Dates: First submitted 2012-05-24; First posted 2012-05-28 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Mental Disorders
Keywords: Lamotrigine; placebo; properties; characteristics
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): To receive the sequence of investigational products in the order of AB where A is cherry lamotrigine ODT and B is cherry placebo.
  Interventions: Drug: Cherry lamotrigine ODT; Drug: Cherry Placebo
- Group 2 (Experimental): To receive the sequence of investigational products in the order of BA where A is cherry lamotrigine ODT and B is cherry placebo.
  Interventions: Drug: Cherry lamotrigine ODT; Drug: Cherry Placebo

INTERVENTIONS:
Drug: Cherry lamotrigine ODT — 25mg, taken orally on one study visit
Drug: Cherry Placebo — Taken orally on one study visit

SUMMARY:
The objective of this sensory analysis study is to determine whether volunteers observe a significant difference in organoleptic properties between lamotrigine (430C78) cherry flavoured orally disintegrating tablets (ODT) and a placebo cherry flavoured orally disintegrating tablet. The aim is to assess the value of the placebo as a marketing aid, whereby physicians and patients may assess the personal acceptability of the organoleptic properties and potential convenience prior to prescription of the ODT formulation.

ELIGIBILITY:
Inclusion Criteria:

A subject will be eligible for inclusion in this study only if all of the following criteria apply:

* Healthy as judged by the responsible physician or designee. No clinically significant abnormality identified on the medical or laboratory evaluation. A subject with a clinical abnormality or laboratory parameters outside the reference range for this age group may be included only if the Investigator and the Medical Monitor considers that the finding will not introduce additional risk factors and will not interfere with the study procedures.
* Volunteer must have a normal sense of taste and smell
* Non-smokers or ex-smokers who have given up smoking for at least 3 months. Subjects currently using oral nicotine replacement therapy will not be recruited for this study.

Exclusion Criteria:

A subject will not be eligible for inclusion in this study if any of the following criteria apply:

* Currently being treated for epilepsy or bipolar disorder
* History of allergic, anaphylactic, hypersensitivity or idiosyncratic reaction(s) to lamotrigine or drugs of a similar type.
* History of sensitivity to any of the following excipients- Mannitol, Crospovidone, Sucralose, Magnesium Stearate, artificial Cherry flavour, Ethylcellulose.
* History of clinically relevant skin rashes.
* History or presence of any medical disorder which in the view of the investigator and GSK Medical Monitor makes the subject unsuitable for the study.
* History of multiple allergies to drugs, chemicals or foods, or a history of a clinically important allergy (e.g. anaphylaxis) to any one substance.
* Currently suffering from perennial rhinitis or seasonal rhinitis, a cold, influenza or any other respiratory illness.
* Has received prescribed or non prescribed medication (including vitamins and herbal remedies) within 7 days prior to the test day which in the opinion of the investigator in consultation if necessary with the GSK Medical Monitor may interfere with the study procedure or compromise safety.
* Currently or recently prescribed any medication which may be affected by lamotrigine including antiepileptics.
* Participation in another sensory analysis study within 30 days preceding the test day.
* Treatment with an investigational drug within 30 days preceding the test day.
* Females with a positive hCG pregnancy test on the test day.
* Abuse of alcohol defined as an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units for men and a weekly intake of greater than14 units or an average daily intake of greater than 2 units for women. [NOTE: 1 unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine]. Subjects must be willing to abstain from alcohol for 24 hours before each visit to the unit for the duration of the study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* The subject has a positive drug/alcohol screen on the test day. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-07-11 (Actual); Primary Completion 2008-07-18 (Actual); Study Completion 2008-07-18 (Actual)

PRIMARY OUTCOMES:
Comparison score of flavor and aftertaste between the active and placebo tablets. | 1 day

SECONDARY OUTCOMES:
Comparison score of mouth feel between the active and placebo tablets | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] This study has not been published in the scientific literature.
- See also: Results for study 111649 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/111649?search=study&study_ids=111649#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111649 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register